CLINICAL TRIAL: NCT01689025
Title: A Randomised, Placebo-controlled, Double-blind, Multiple-dose, Dose-escalation Trial Investigating the Safety and Tolerability of NNC0114-0006 in Subjects With Systemic Lupus Erythematosus
Brief Title: An Investigation of Safety and Tolerability of NNC0114-0006 in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8828-4002; 2011-005699-41 (EudraCT Number); U1111-1125-9646 (Other: WHO)
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Inflammation; Systemic Lupus Erythematosus
MeSH Terms: conditions — Inflammation; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0114-0006 (Experimental)
  Interventions: Drug: NNC0114-0006
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0006 — Administered subcutaneously (s.c., under the skin) every second week to a total of four doses.
  Arms: NNC0114-0006
Drug: placebo — Administered subcutaneously (s.c., under the skin) every second week to a total of four doses.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of the trial is to investigate the safety and tolerability of NNC0114-0006 in subjects with systemic lupus erythematosus (SLE) concomitantly treated with stable background therapies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (not pregnant and not nursing)
* Subjects with SLE meeting the American College of Rheumatology (ACR) criteria, with a disease duration of at least 6 months
* Subjects with clinically active SLE defined as a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score of at least 6 and positive for antinuclear antibody (ANA) and/or Anti-double-stranded DNA antibody (anti-dsDNA)
* If taken, background medication must be stable

Exclusion Criteria:

* Presence or history of active lupus nephritis (LN) within the last 4 months or active central nervous system (CNS) disease within the last 12 months
* Body mass index (BMI) below 18 kg/m^2 or above 38 kg/m^2

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first administration of the trial product and up to week 26

SECONDARY OUTCOMES:
PK endpoint from serum NNC0114-0006: Terminal elimination half-life (t½) | After the last dosing (Week 6)
PK endpoint from serum NNC0114-0006: Accumulation based on the concentration | 2 weeks after the first (week 2) and the last dose (week 8)
Change in serum levels of total IL-21 (Interleukin-21) | Week 0, week 26
Change in disease activity (SELENA-SLEDAI) | Week 0, week 12
Change in corticosteroid usage | Week 0, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- United States (2):
  - Novo Nordisk Clinical Trial Call Center, La Jolla, California
  - Novo Nordisk Clinical Trial Call Center, Houston, Texas
- Szeged, Hungary
- Poznan, Poland
- Belgrade, Serbia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com